CLINICAL TRIAL: NCT02455167
Title: Reversal of Hepatic Impairment by Achieving Sustained Virologic Response (SVR) With 12 Weeks of Simeprevir(SMV)/Sofosbuvir(SOF)/Ribavirin(RBV) in Patients With Hepatitis C Virus (HCV) Genotype 1 Infection and Early Decompensation of Cirrhosis (MELD 10 or Less)
Brief Title: Reversal of Hepatic Impairment in Patients With Hepatitis C Virus (HCV) and Early Decompensation of Cirrhosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped due to low accrual and availability of other treatment options
Sponsor: University of Colorado, Denver (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-0919; UL1TR001082 (NIH)
Record Dates: First submitted 2015-04-21; First posted 2015-05-27 (Estimated); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis C
Keywords: HCV; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HCV positive group (Experimental): A single arm study of 'Simeprivir (SMV), Sofosbuvir (SOF) and Ribavirin (RBV) in an HCV positive population.
  Interventions: Drug: Simeprivir (SMV); Drug: Sofosbuvir (SOF); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Simeprivir (SMV) — Experimental Single arm study. All participants will get the same treatment.
  Other Names: Olysio (Simeprivir);
Drug: Sofosbuvir (SOF) — Experimental Single arm study. All participants will get the same treatment.
  Other Names: Solvaldi (Sofosbuvir);
Drug: Ribavirin (RBV) — Experimental Single arm study. All participants will get the same treatment.
  Other Names: Virazole (Ribavirin);

SUMMARY:
1. Achieve sustained virologic response (SVR) in patients infected with HCV genotype 1, cirrhosis, and early clinical decompensation using 12 weeks of Olysio/Sovaldi/Ribavirin (or known as: Simeprevir(SMV)/Sofosbuvir(SOF)/Ribavirin (RBV).
2. Hepatic improvement during and after Simeprevir(SMV)/Sofosbuvir(SOF)/Ribavirin(RBV) treatment using a new test of liver function, HepQuant-SHUNT.

DETAILED DESCRIPTION:
The proposed study will quantify hepatic improvement and antiviral efficacy of the open-label interferon-free combination of 12 weeks of simeprevir (SMV, Simeprevir), sofosbuvir (SOF, Sofosbuvir), and ribavirin (RBV) in patients with HCV genotype 1 infection and early decompensation of cirrhosis. Early decompensation is defined by clinical complications or laboratory deterioration but with a model for end-stage liver disease (MELD) score of 10 or less.

The primary objective of this trial is determination of hepatic functional improvement as measured by the HepQuant (HQ) test during and after Simeprevir(SMV)/Sofosbuvir(SOF)/Ribavirin(RBV). Standard laboratory tests, clinical models (MELD, CTP), liver biopsy, hepatic venous pressure gradient (HVPG), and other imaging tests are insensitive, invasive, or nonspecific.

They may not adequately assess the liver's improvement after viral eradication. In contrast, HepQuant (HQ) tests (Systemic Hepatic Filtration Rate (HFR), Portal HFR, SHUNT,single point cholate concentration (STAT), and DSI) are noninvasive, sensitive, specific, and target an endogenous function, the hepatic uptake of cholate. HQ tests uses serum sampling over a time period of up to 90 minutes to quantify the systemic circulation, portal circulation, and portal-systemic shunt and to derive a disease severity index (DSI) in intact human subjects. The primary endpoint in this treatment trial will be improvement in hepatic function measured by HepQuant (HQ) tests that occurs during and after successful Simeprevir(SMV)/Sofosbuvir(SOF)/Ribavirin(RBV).

ELIGIBILITY:
Inclusion Criteria:

1. HCV genotype 1 infection (all subtypes and Q80K a type of mutation are allowed), and have been approved by a third party payer for the FDA-approved combination of sofosbuvir (SOF) plus ribavirin. The study drug, simeprevir (SMV)
2. Biopsy proven cirrhosis, or clinical cirrhosis with APRI (AST to Platelet Ratio Index to determine clinical cirrhosis)> 2, Fibrotest > 0.75, or Fibroscan > 12.5 Results Stiffness (kPa).
3. MELD 10 or less
4. Expected survival without liver transplantation of >1 year
5. Patients with Hepatocellular carcinoma (HCC) are included as long as disease MELD is 10 or less, and anticipated time to transplant is >1 year. An example, might be a patient with a subcentimeter HCC who is undergoing serial imaging to document tumor growth to tumor diameter >2 cm prior to listing for transplantation (in order to secure MELD exception). In this case, there could be a time lapse of 3 months or more while monitoring tumor growth, and a further time lapse of 9 months or more until the time of transplantation.
6. Patients with TIPS or Portal Vein Thrombosis may be included. -

Exclusion Criteria:

1. Inability to provide informed consent
2. Known hypersensitivity or serious adverse reaction to any of the study drugs
3. Age <18 or >80 years
4. Pregnancy as determined by subject reporting and urine dipstick testing at screening.
5. Other underlying chronic liver disease - examples that would exclude a patient from participating include but are not limited to nonalcoholic liver disease, alcoholic liver disease, hepatitis B, hemochromatosis, and autoimmune liver disease.
6. Serious other underlying medical condition - examples include but are not limited to unstable cardiovascular, coronary, or pulmonary disease including right and left sided heart failure, active malignancy other than HCC, or serious infection.
7. Estimated creatinine clearance < 30 mL min-1 1.73 m2 surface area (BSA)
8. Hemoglobin <10 g/dL
9. Neutrophils <500 /μL
10. Platelets <50,000 /μL
11. Bilirubin >4 mg/dL
12. Albumin < 2.8 g/dL
13. Blood Clotting: International Normalised Ratio (INR) > 2
14. MELD >10
15. Child-Turcotte-Pugh class B or C; or, CTP score >7
16. Conditions that would affect the absorption of orally administered cholate used in the HepQuant® test - such as, extensive intestinal resection, diabetic gastroparesis, and ileal disease or resection.
17. Concomitant use of both beta-blocker and ACE inhibitor
18. Subjects taking any other medications with significant drug drug interactions related to the study medications (sofosbuvir, simeprevir, or ribavirin) who cannot discontinue or substitute that medication, will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-05; Primary Completion 2016-07-18 (Actual); Study Completion 2016-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Wieland, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver (Leprino Building), Denver, Colorado, United States

REFERENCES:
- [Result] Everson GT, Martucci MA, Shiffman ML, Sterling RK, Morgan TR, Hoefs JC; HALT-C trial group. Portal-systemic shunting in patients with fibrosis or cirrhosis due to chronic hepatitis C: the minimal model for measuring cholate clearances and shunt. Aliment Pharmacol Ther. 2007 Aug 1;26(3):401-10. doi: 10.1111/j.1365-2036.2007.03389.x. PMID 17635375
- [Result] Everson GT, Shiffman ML, Morgan TR, Hoefs JC, Sterling RK, Wagner DA, Kulig CC, Curto TM, Wright EC; Halt-C Trial Group. The spectrum of hepatic functional impairment in compensated chronic hepatitis C: results from the Hepatitis C Anti-viral Long-term Treatment against Cirrhosis Trial. Aliment Pharmacol Ther. 2008 May;27(9):798-809. doi: 10.1111/j.1365-2036.2008.03639.x. Epub 2008 Feb 7. PMID 18266997
- [Result] Everson GT, Shiffman ML, Hoefs JC, Morgan TR, Sterling RK, Wagner DA, Desanto JL, Curto TM, Wright EC; HALT-C Trial Group. Quantitative tests of liver function measure hepatic improvement after sustained virological response: results from the HALT-C trial. Aliment Pharmacol Ther. 2009 Mar 1;29(5):589-601. doi: 10.1111/j.1365-2036.2008.03908.x. Epub 2008 Dec 1. PMID 19053983
- [Result] Everson GT. Hepatic cysts in autosomal dominant polycystic kidney disease. Am J Kidney Dis. 1993 Oct;22(4):520-5. doi: 10.1016/s0272-6386(12)80923-1. No abstract available. PMID 8213790
- [Result] Shrestha R, McKinley C, Showalter R, Wilner K, Marsano L, Vivian B, Everson GT. Quantitative liver function tests define the functional severity of liver disease in early-stage cirrhosis. Liver Transpl Surg. 1997 Mar;3(2):166-73. doi: 10.1002/lt.500030210. PMID 9346731
- [Result] Shaheen AA, Wan AF, Myers RP. FibroTest and FibroScan for the prediction of hepatitis C-related fibrosis: a systematic review of diagnostic test accuracy. Am J Gastroenterol. 2007 Nov;102(11):2589-600. doi: 10.1111/j.1572-0241.2007.01466.x. Epub 2007 Sep 10. PMID 17850410
- [Result] Tripodi A, Caldwell SH, Hoffman M, Trotter JF, Sanyal AJ. Review article: the prothrombin time test as a measure of bleeding risk and prognosis in liver disease. Aliment Pharmacol Ther. 2007 Jul 15;26(2):141-8. doi: 10.1111/j.1365-2036.2007.03369.x. PMID 17593061

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants screen-failed after enrollment.
Period: Overall Study
Arm/Group | HCV Positive Group
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HCV Positive Group
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 57 [40 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: The Sustained Virologic Response (SVR) in Patients Infected With HCV Genotype 1, Cirrhosis, and Early Clinical Decompensation
Description: Number of participants who cleared Hepatitis C (HCV) after 12 weeks was collected (HCV RNA level was "Not Detected".
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | HCV Positive Group
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Hepatic Improvement During and After Simeprevir(SMV)/Sofosbuvir(SOF)/Ribavirin(RBV) Treatment Using a New Test of Liver Function, HepQuant-SHUNT: Baseline
Description: Liver function as assessed via MELD score. The Model For End-Stage Liver Disease (MELD) score assesses the severity of patient liver disease. Possible scores range from 6 to 40, with higher scores indicating more severe liver disease and a worse outcome.
Time Frame: Baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | HCV Positive Group
Number analyzed (Participants) | 4
score on a scale | 8 [7 to 10]

3. Primary Outcome: Hepatic Improvement During and After Simeprevir(SMV)/Sofosbuvir(SOF)/Ribavirin(RBV) Treatment Using a New Test of Liver Function, HepQuant-SHUNT: 12 Weeks
Description: as for outcome 2
Time Frame: 12 Weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | HCV Positive Group
Number analyzed (Participants) | 4
score on a scale | 7.25 [7 to 8]

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | HCV Positive Group
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HCV Positive Group (N=4)
Protocol deviation (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes